CLINICAL TRIAL: NCT00005384
Title: Diet/Activity of Mexican American and Anglo Children
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4289; R01HL052449 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To perform a follow-up study of physical activity and dietary behaviors and their determinants in 10- to 11-year-old Anglo and Mexican-American children from low- and middle-socioeconomic status (SES) families who were studied initially when they were 4 to 7 years old.

DETAILED DESCRIPTION:
BACKGROUND:

It is well documented that the roots of cardiovascular diseases (CVD) are evident in childhood, and elevated levels of serum lipids, blood pressure and body fat are common in childhood. These risk factors are, in turn, related to childhood dietary and physical activity habits. To understand the early development of CVD, it is therefore important to study factors that influence diet and physical activity behaviors in children. Most studies concerned with the determinants of diet and physical activity in children are cross-sectional, limiting their utility for improving understanding of the development of these key health behaviors.

The study allowed prospective analyses of the behaviors over a significant portion of the prepubertal age range. Knowledge of the determinants, stability, and relationships of childhood dietary and physical activity behaviors to physiologic risk variables could be useful for setting priorities and designing public health interventions for the next generations of youth.

The major contribution of this San Diego SCAN study was in the longitudinal analysis of dietary and physical activity behaviors in children. The follow-up assessment of the 10-to 11-year-old cohort and their mothers produced data that substantially improved understanding of the determinants and tracking of children's dietary and physical activity behaviors, as well as their relations to CVD risk factors.

DESIGN NARRATIVE:

Selection of subjects studied was based on social learning/cognitive theory, which states that behaviors are a function of personal and environmental factors. The specific aims of the study were as follows: 1) To study the determinants of physical activity and dietary intake of fat, sodium, and calories, and changes in these behaviors in children from ages 4 to 10-11. 2) To determine the relationships between diet and physical activity practices and physiologic indicators of risk, such as blood pressure, adiposity, body mass, and serum lipoproteins at ages 4 to 10-11. 3) To describe the time trends and the degree of tracking of physical activity habits and nutritional intake of fat, sodium, and calories in children from ages 4 to 10-11. The study was renewed in 1999.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1995-01; Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Nader — University of California, San Diego

REFERENCES:
- [Background] Reaven P, Nader PR, Berry C, Hoy T. Cardiovascular disease insulin risk in Mexican-American and Anglo-American children and mothers. Pediatrics. 1998 Apr;101(4):E12. doi: 10.1542/peds.101.4.e12. PMID 9521978
- [Background] Masu R, Sallis JF, Berry CC, Broyles SL, Elder JP, Nader PR. The relationship between health beliefs and behaviors and dietary intake in early adolescence. J Am Diet Assoc. 2002 Mar;102(3):421-4. doi: 10.1016/s0002-8223(02)90099-4. No abstract available. PMID 11902380
- [Background] Sallis JF, Greenlee L, McKenzie TL, Broyles SL, Zive MM, Berry CC, Brennan J, Nader PR. Changes and tracking of physical activity across seven years in Mexican-American and European-American mothers. Women Health. 2001;34(4):1-14. doi: 10.1300/J013v34n04_01. PMID 11785854
- [Background] Frank GC, Nader PR, Zive MM, Broyles SL, Brennan JJ. Retaining school children and families in community research: lessons from the Study of Children's Activity and Nutrition (SCAN). J Sch Health. 2003 Feb;73(2):51-7. doi: 10.1111/j.1746-1561.2003.tb03571.x. PMID 12643019